CLINICAL TRIAL: NCT03167008
Title: Correlation Between the Level of Vitamin D and Semen Parameters
Brief Title: Vitamin D Level vs Semen Parameters
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, kh, Principal Investigator, Assiut University
Other Study IDs: VDSP
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- idiopathic male infertility: * total of 30 male patients with idiopathic male infertility.
  * Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010).
  * blood samples will be taken &the following will be done Serum vitamin D level ,Serum calcium level ,Serum testosterone level ,luteinizing hormone (LH), and follicle-stimulating hormone (FSH), will be measured.
  Interventions: Diagnostic Test: semen sample; Diagnostic Test: blood sample
- fertile male group: * total of 30 fertile male (as control)
  * Semen samples will be collected,Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010).
  * blood samples will be taken &the following will be done Serum vitamin D level ,Serum calcium level ,Serum testosterone level ,luteinizing hormone (LH), and follicle-stimulating hormone (FSH), will be measured.
  Interventions: Diagnostic Test: semen sample; Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: semen sample — -Semen samples will be collected from all patients Semen analysis will be examined after 2-5 days of sexual abstinence based on World Health Organization (WHO) (2010)
Diagnostic Test: blood sample — blood samples will be taken &the following will be done Serum vitamin D level ,Serum calcium level ,Serum testosterone level ,luteinizing hormone (LH), and follicle-stimulating hormone (FSH), will be measured

SUMMARY:
* Infertility is defined as the inability of a sexually active couple to conceive after 1 year of regular intercourse without contraception, affects approximately 15% of couples, and male factors are the cause in 20% -50% of cases.
* Infertility of unknown origin is classified into idiopathic male infertility and unexplained male infertility according to semen quality.

DETAILED DESCRIPTION:
-Idiopathic male infertility is known as idiopathic oligoasthenoteratozoospermia, which indicates that the men have an unexplained reduction of semen quality.

In contrast, unexplained male infertility is defined as infertility of unknown origin with normal sperm parameters.

Furthermore, optimal strategies for treating idiopathic male infertility have also remained unclear.

* Data from studies in humans suggest that vitamin D receptors are present in testis, epididymis, prostate and seminal vesicles. The level of expression varies, being higher in epididymis and seminal vesicles.
* Vitamin D receptors expression was also evident in Leydig cells, as well as in normal and abnormal sperm, with the acrosomal region and the neck being the sites with the most abundant messenger ribonucleic acid expression.
* The 1,25(OH)2 D3 molecule increases intracellular calcium concentrations, sperm motility and acrosin activity, and reduces triglyceride content in sperm, actions that significantly contribute to fertilising capacity within the female reproductive tract.

ELIGIBILITY:
Inclusion Criteria:

* infertile male patients without any detectable cause with normal clinical examination and abnormal semen parameters.

Exclusion Criteria:

* Cases with known etiology or apparent physical finding ,leukocytospermia, diminished testicular volume ,varicocele or an abnormal hormonal profile.
* couples with combined male and female factor will be excluded.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: total of 30 male patients with idiopathic male infertility and other 30 fertile male (as control) will be randomly recruited from the outpatient andrology clinic of the department at Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
correlation between vitamin D level and semen parameters | baseline

CONTACTS AND LOCATIONS:
Overall Officials: MAKhair, Principal Investigator — Assiut University

REFERENCES:
- [Background] Irvine DS. Epidemiology and aetiology of male infertility. Hum Reprod. 1998 Apr;13 Suppl 1:33-44. doi: 10.1093/humrep/13.suppl_1.33. PMID 9663768
- [Background] Gnoth C, Godehardt E, Frank-Herrmann P, Friol K, Tigges J, Freundl G. Definition and prevalence of subfertility and infertility. Hum Reprod. 2005 May;20(5):1144-7. doi: 10.1093/humrep/deh870. Epub 2005 Mar 31. PMID 15802321
- [Background] Ko EY, Siddiqi K, Brannigan RE, Sabanegh ES Jr. Empirical medical therapy for idiopathic male infertility: a survey of the American Urological Association. J Urol. 2012 Mar;187(3):973-8. doi: 10.1016/j.juro.2011.10.137. Epub 2012 Jan 20. PMID 22264467
- [Background] Blomberg Jensen M, Nielsen JE, Jorgensen A, Rajpert-De Meyts E, Kristensen DM, Jorgensen N, Skakkebaek NE, Juul A, Leffers H. Vitamin D receptor and vitamin D metabolizing enzymes are expressed in the human male reproductive tract. Hum Reprod. 2010 May;25(5):1303-11. doi: 10.1093/humrep/deq024. Epub 2010 Feb 18. PMID 20172873
- [Background] Walters MR. 1,25-dihydroxyvitamin D3 receptors in the seminiferous tubules of the rat testis increase at puberty. Endocrinology. 1984 Jun;114(6):2167-74. doi: 10.1210/endo-114-6-2167. PMID 6327237